CLINICAL TRIAL: NCT02908126
Title: Compare Efficacy of Oxytocin Administrations on Postpartum Uterine Contractility
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No approval CA (MPA) of protocol amendment
Sponsor: Oxytone Bioscience BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OXB-002
Record Dates: First submitted 2016-09-16; First posted 2016-09-20 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Post Partum Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin intravenous (Experimental): single dose of intravenous (IV) oxytocin
  Interventions: Drug: Oxytocin
- Oxytocin tablet (Experimental): single dose of oxytocin tablet
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin drug

SUMMARY:
This is a Phase I open-label, parallel-group clinical study in healthy term pregnant females undergoing a caesarean section. Two administrations of oxytocin will be tested, after which uterine contractility will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, term pregnant female with a gestational age of 37-42 weeks (singleton)
* Undergoing a planned primary and uncomplicated caesarean section (CS) for their first born under regional anaesthesia
* Aged between 18 and 40 years (both inclusive)
* Ability to communicate well with the Investigator and to comply with the requirements of the entire study
* Willing to give informed consent in writing.

Exclusion Criteria:

* Being obese with BMI ≥35 before pregnancy
* History of, or existing thromboembolic, cardiovascular or cerebrovascular disorder
* History of cervical cancer
* History of severe infection of the uterus
* Previous surgery of the cervix or uterus or any other (previous) condition that could interfere with the measurement of uterine contractility
* Any clinically significant abnormality following review of medical history, laboratory result and physical examination at screening as judged by the Investigator
* Conditions or disorders that might affect the absorption, distribution, metabolism or excretion of any of the study medication
* Contraindications for oxytocin use
* Hypersensitivity to the active substances or to any of the excipients of the investigational product (test product or comparator drug)
* Present use or use within 30 days before the start of the study medication of one or more of the following medications: antihypertensive drugs, anti-coagulant therapy, medication that could affect myometrial contractility, sex steroids, prostaglandins and its analogues, inhalation anaesthetics, vasoconstrictors/sympathomimetics and caudal anaesthetics, vasopressin-like drugs
* Administration of any other investigational drug within 3 months before first dosing
* Tobacco use (smoking or snuffing), currently or within the last 6 months before screening

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Uterine contractility: area under the curve (AUC) | 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institute, Danderyd hospital,Dept of Obstetrics and Gynecology, Stockholm, Sweden